CLINICAL TRIAL: NCT00533975
Title: A Prospective Study of a New Immunochemical Fecal Occult Blood Test in U.S. Veteran Patients Undergoing Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of California, San Diego (Other)
Other Study IDs: 071015
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-06

CONDITIONS: Colon Cancer
Keywords: Colon Cancer screening; immunofecal occult blood test; colonoscopy; diagnostic validity
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of our study is to evaluate the diagnostic validity of a new immunofecal occult blood test (IFOBT) (Teco Diagnostics) in U.S. veterans and to compare it with the guaiac based FOBT.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer in men and women in the United States with an estimated 147,000 new cases and more than 56,000 deaths each year. Early detection of colon cancer and removal of precancerous adenomatous polyps have been shown to reduce its morbidity, mortality and incidence. There are several recommended CRC screening tests, including fecal occult blood test (FOBT), flexible sigmoidoscopy, air-contrast barium enema, and colonoscopy. In the VA, FOBT is the predominant screening test for CRC. Numerous randomized controlled trials have established the efficacy of FOBT in CRC screening. Its advantages include privacy, noninvasiveness, and cost-effectiveness. Use of guaiac-based testing, however, is hampered by low patient compliance, sensitivity, specificity, and positive predictive value. The poor patient compliance, and low specificity and positive predictive value, may be related to the testing procedure. For example, dietary and medication restrictions are recommended to decrease false-negative and false-positive tests. Such restrictions may impede patient compliance. Recently, several studies have evaluated the effectiveness immunochemical-based testing as a potential alternative, with reportedly better compliance, sensitivity, and specificity than guaiac-based tests. The purpose of our study is to evaluate the diagnostic validity of a new IFOBT (Teco Diagnostics) in U.S. veterans and to compare it with the guaiac based FOBT.

ELIGIBILITY:
Inclusion Criteria:

* Patients (men or women) that are >18 years of age undergoing colonoscopy for a variety of indications (bleeding, diarrhea, weight loss, anemia, abdominal pain, etc)

Exclusion Criteria:

* concurrent hospitalization
* visible rectal bleeding
* known diagnosis of inflammatory bowel disease
* hematuria
* menstruation at the time of obtaining a stool specimen and performing the tests
* inability to prepare the 3 different IFOBT or 3 different FOBT kits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-09; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel B Ho, M.D., Principal Investigator — UCSD, VA San Diego
Locations (1):
- Veteran Affairs Medical Center San Diego, San Diego, California, United States